CLINICAL TRIAL: NCT04088513
Title: A Randomized, Double-blind, Active-Controlled Trial Comparing the Safety and Efficacy of Aspirin Versus Clopidogrel in Stroke Patients With Glucose-6-phosphate Dehydrogenase Deficiency
Brief Title: Safety and Efficacy of Aspirin in Stroke Patients With Glucose-6-phosphate Dehydrogenase Deficiency (SAST)
Acronym: SAST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinsheng Zeng, MD, PhD, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAST; 2018001 (Other Grant/Funding Number: Sun Yat-Sen University)
Record Dates: First submitted 2019-09-08; First posted 2019-09-12 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: G6PD Deficiency; Stroke
Keywords: G6PD Deficiency; Acute ischemic stroke; Aspirin; Hemolysis; Clopidogrel; Anti-platelet therapy
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency; Stroke; Ischemic Stroke; Hemolysis | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Drugs:Aspirin
  Interventions: Drug: Aspirin
- Clopidogrel (Active Comparator): Drugs:Clopidogrel
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin — This group will receive a 100 mg/day aspirin plus clopidogrel placebo for 90 days.
  Other Names: Acetylsalicylic acid
  Arms: Aspirin
Drug: Clopidogrel — This group will receive a 75 mg/day clopidogrel plus aspirin placebo for 90 days.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
Aspirin was reported to induce hemolysis in patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency on some occasions, while still widely uesd for stroke prevention. The SAST trial is designed to evaluate the safety and efficacy of aspirin in patients this enzyme disorder.The primary purpose of the trial is to evaluate the hemolytic effects of a 3-month regimen of aspirin 100mg/d versus a 3-month regimen of clopidogrel 75mg/d.

DETAILED DESCRIPTION:
This SAST trial is a prospective, multicenter, randomized, double-blind trial.440 acute ischemic stroke (AIS) patients with G6PD deficiency will be randomized to receive a 3-month regimen of aspirin 100mg/d or clopidogrel 75mg/d. The primary end point is the proportion of protocol-defined hemolysis at 90 days. Protocol-defined hemolysis is defined as one or more of the following conditions: a) Hemoglobin level declined ≥2.5 g/dL from baseline, meanwhile ruling out bleeding events. b) Hemoglobin level declined ≥25% from baseline, meanwhile ruling out bleeding events. c) Clinically relevant hemolytic events, could manifested as fatigue, back pain, anemia, dark urine and jaundice. The study consists of five visits including the day of randomization, day 4, day10±3days, day27±3days, day90±7days.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥40 years(no upper limit)
2. Acute ischemic stroke within 14 days of symptoms onset;
3. Glucose-6-phosphate dehydrogenase deficiency screened in G6PD enzyme activity
4. Had not received aspirin 7 days prior to randomization
5. Informed consent signed

Exclusion Criteria:

1. Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other non-ischemic brain disease, base on head CT or MRI
2. Concomitant infections at the time of randomization
3. mRS>2 prior to the presenting stroke
4. Hemoglobin<10 g/dL prior to randomization
5. Received intravenous thrombolytic therapy or neurointervention treatment before randomization
6. Clear indication for anticoagulation (presumed cardioembolism, eg, atrial fibrillation, prosthetic cardiac valves or suspected endocarditis)
7. Clear indication for dual antiplatelet therapy (eg, minor stroke in 24h (NIHSS ≤3) or endovascular therapy for the indexed event)
8. Anticipated concomitant antiplatelets other than aspirin or clopidogrel (eg, GPIIb/IIIa inhibitors, ticlopidine, prasugrel, dipyridamole, ozagrel, cilostazol, ticagrelor) and other antithrombotic agents with antiplatelet effects, including traditional/herbal medicine agents.
9. Anticipated concomitant therapy with long-term (>7 days) NSAIDs affecting platelet function
10. Contraindication to clopidogrel or aspirin (1)Known allergic reactions (2)Severe hepatic or renal dysfunction (Severe hepatic dysfunction is defined as serum ALT or AST >2 times the upper limit of the normal group；Severe renal dysfunction is defined as serum creatinine > 1.5 times the upper limit of the normal group) (3)Severe cardiac failure（NYHA class Ⅲ or Ⅳ) (4)Asthma (5)Any history of Hemostatic disorder or systemic bleeding (6)Any history of thrombocytopenia or neutropenia (7)Any history of drug-induced hematologic or hepatic insufficiency (8)Low white blood cell (<2×10^9/L) or platelet count (<100×10^9/L)
11. Any history of thalassemia, autoimmune hemolytic disease, aplastic anemia or other severe hematologic diseases
12. Anticipated concomitant therapy with other contraindicated drugs for G6PD deficiency
13. Severe dysphagia to unable swallow the drugs
14. Concomitant infections and need for antimicrobial therapy
15. Intracranial hemorrhage or gastrointestinal bleed within 3 months, or major surgery within 30 days
16. Stomach tumor or any other malignant tumor
17. Planed surgery or interventional treatment that may affect the study procedure
18. Severe non-cardiovascular comorbidity with life expectancy <3 m
19. Female who is pregnant or lactating
20. Currently receiving an investigational drug or device
21. Inability to understand and/or comply with study procedures due to psychosis, cognition impairment or emotion disturbance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of protocol-defined hemolysis. | 90±5 days.
  Protocol-defined hemolysis is defined as one or more of the following conditions: a) Hemoglobin level declined ≥2.5 g/dL from baseline, meanwhile ruling out bleeding events. b) Hemoglobin level declined ≥25% from baseline, meanwhile ruling out bleeding events. c) Clinically relevant hemolytic events, could manifested as fatigue, back pain, anemia, dark urine and jaundice, adjudicated by the adjudication committee ultimately.

SECONDARY OUTCOMES:
Change in hemoglobin. | 4 days,10±3 days,27±3 days and 90±5 days.
Change in reticulocyte. | 4 days,10±3 days,27±3 days and 90±5 days.
Change in unconjugated bilirubin and total bilirubin. | 4 days,10±3 days,27±3 days and 90±5 days.
Change in lactic dehydrogenase. | 4 days,10±3 days,27±3 days and 90±5 days.
Proportion of major bleed (GUSTO deﬁnition). | 90±5 days.
Overall mortality. | 90±5 days.
Proportion of new clinical vascular events, deﬁned as the composite of stroke, transient ischemic attack (TIA), myocardial infarction and vascular death. | 90±5 days.
Proportion of functional independence defined as modified Rankin Scale score 0-2. | 90±5 days.
  Modified Rankin Scale score ranges from 0 to 6, and lower score means more functional independence.
Proportion of functional independence defined as Barthel Index 95-100. | 90±5 days.
  Barthel Index ranges from 0 to 100, and higher score means more functional independence.
Change in National Institutes of Health Stroke Scale | 90±5 days.
  National Institutes of Health Stroke Scale ranges from 0 to 42, and higher scores indicate more severe neurologic deficits.
Health related quality of life, assessed by EuroQoL-5 Dimensions questionnaire | 90±5 days.
  EuroQoL-5 Dimensions questionnaire contains utility index score and visual analogue scale. Utility index score ranges from 0 to 1, and visual analogue scale ranges from 0 to 100. Higher scores indicate more healthy quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsheng Zeng, MD,PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (19):
- China (19):
  - Longyan First Hospital, Longyan, Fujian
  - Sanming First Hospital, Sanming, Fujian
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Jieyang Municipal People's Hospital, Jieyang, Guangdong
  - Meizhou City People's Hospital, Meizhou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - Yunfu People's Hospital, Yunfu, Guangdong
  - People's Hospital of Baise, Baise City, Guangxi
  - The Forth Affiliated Hospital of Guangxi Medical Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical Hospital, Nanning, Guangxi
  - Beiliu People's Hospital, Yulin, Guangxi
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Fengcheng People's Hospital, Fengcheng, Jiangxi
  - Ganzhou Municipal Hospital, Ganzhou, Jiangxi
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Ganzhou People' Hospital, Ganzhou, Jiangxi
  - The Forth Affiliated Hospital of Nanchang University, Nanchang, Jiangxi